CLINICAL TRIAL: NCT06540716
Title: Inspire Singapore Study: Confirmation of Therapy Performance
Brief Title: Inspire Singapore Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-001
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea; OSA; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hypoglossal nerve stimulation (Other)
  Interventions: Device: Inspire System

INTERVENTIONS:
Device: Inspire System — Hypoglossal nerve stimulation therapy will be activated at approximately 1 month post-implant.

SUMMARY:
Prospective, multicenter, open-label study designed to confirm device performance of Inspire system in Singapore.

DETAILED DESCRIPTION:
Patients who meet study eligibility criteria will be implanted with an Inspire system and followed for 6 months post-therapy-activation. Study subjects will undergo in-lab sleep studies to confirm inspiratory overlap (1st PSG, after therapy activation), titrate the therapy (2nd PSG, at 3 months post-activation) and confirm therapy performance (3rd PSG, at 6 months post-activation). Symptoms and quality of life (assessed by ESS and FOSQ), therapy adherence, and adverse events will also be collected and reported.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of moderate to severe OSA (AHI 15-65)
* Failure of, or intolerance to CPAP

Main Exclusion Criteria:

* Central + mixed apneas > 25% of total AHI
* Presence of complete concentric collapse (CCC)
* Compromised neurological control of the upper airway.

Other eligibility criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Inspiratory Overlap | 0-3 months post-therapy activation
  Percentage (%) of inspiratory overlap as measured by polysomnography (PSG)

SECONDARY OUTCOMES:
Therapy Effectiveness | 6 months post-therapy activation
  Change in Apnea-Hypopnea Index (AHI)
Symptom Reduction | 6 months post-therapy activation
  Mean Epworth Sleepiness Scale (ESS) Score of less than 10. ESS scores range from 0-24 with a score of less than 10 indicating normalized daytime sleepiness.

OTHER OUTCOMES:
Rate of Adverse Events | 6 months post-therapy activation
  Report of procedure/device/therapy-related adverse events
Therapy Adherence | 6 months post-therapy activation
  Mean therapy use (hours per day)
Functional Outcomes of Sleep Questionnaire (FOSQ) Score | 6 months post-therapy activation
  Changes in Functional Outcomes of Sleep Questionnaire (FOSQ). Total score range 5-20, with higher scores indicating better functional status.
Inspiratory Overlap | 6 months post-therapy activation
  Percentage (%) of inspiratory overlap as measured by polysomnography (PSG)

CONTACTS AND LOCATIONS:
Overall Officials: Toh Song Tar, MD, Principal Investigator — Singapore General Hospital
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.